CLINICAL TRIAL: NCT03988036
Title: A Prospective, Multicenter, Open Label, Neoadjuvant Phase II Single Arm Study With Pembrolizumab in Combination With Dual Anti-HER2 Blockade With Trastuzumab and Pertuzumab in Early Breast Cancer Patients With Molecular HER2-enriched Intrinsic Subtype
Brief Title: A Study With Pembrolizumab in Combination With Dual Anti-HER2 Blockade With Trastuzumab and Pertuzumab in Early Breast Cancer Patients With Molecular HER2-enriched Intrinsic Subtype (Keyriched-1)
Acronym: Keyriched-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); NanoString Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM09; 2018-003996-37 (EudraCT Number)
Record Dates: First submitted 2019-03-07; First posted 2019-06-17 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: HR positive; HER2 negative; Early breast cancer; Neoadjuvant; Anti-HER2 therapy; Pertuzumab; Trastuzumab; Pembrolizumab; Immune checkpoint inhibitor; PD-1; PDL-1; PAM50; Phase 2
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; Trastuzumab; pertuzumab

STUDY DESIGN:
Intervention Model Description: A multicenter, interventional, prospective, single arm, open label, neoadjuvant phase II trial evaluating the pathological complete response (pCR) rate induced by pembrolizumab in combination with the dual anti-HER2 blockade consisting of trastuzumab biosimilar and pertuzumab in early breast cancer patients with molecular HER2-enriched intrinsic subtype tested by PAM50.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HER2-enriched (Experimental): Trial treatment is defined as neoadjuvant therapy only. The Investigational Medicinal Products (IMPs) are pembrolizumab, trastuzumab biosimilar and pertuzumab.
  * Trastuzumab Biosimilar (Trazimera®) - Investigational Medicinal Product
    * Loading dose: 8 mg/kg bodyweight at initial administration infusion over 90 min; monitor patient for at least 6 h afterwards.
    * Maintenance dose: 6 mg/kg bodyweight, over 30-90 min; monitor patient for 2 h afterwards.
    * Route: Intravenous infusion.
    * Schedule: Every 3 weeks during the neoadjuvant phase.
  * Pertuzumab (Perjeta®) - Investigational Medicinal Product
    * Loading dose: 840 mg, initial administration.
    * Maintenance dose: 420 mg.
    * Route: Intravenous infusion.
    * Schedule: Every 3 weeks during the neoadjuvant phase.
  * Pembrolizumab (Keytruda®) - Investigational Medicinal Product
    * Dose: 200 mg.
    * Route: Intravenous infusion.
    * Schedule: Every 3 weeks during the neoadjuvant phase.
  Interventions: Drug: Pembrolizumab; Drug: Trastuzumab Biosimilar ABP 980; Drug: Pertuzumab

INTERVENTIONS:
Drug: Pembrolizumab — Intravenous infusion; 200 mg; every 3 weeks
  Other Names: Keytruda®
Drug: Trastuzumab Biosimilar ABP 980 — Intravenous infusion; 8 mg/kg loading dose, thereafter 6 mg/kg; every 3 weeks
  Other Names: Trazimera®
Drug: Pertuzumab — Intravenous infusion; 840 mg/kg loading dose, thereafter 420 mg/kg; every 3 weeks
  Other Names: Perjeta®

SUMMARY:
Keyriched-1 is a multicenter, interventional, prospective, single arm, open label, neoadjuvant phase II trial evaluating the pathological complete response (pCR) rate induced by pembrolizumab in combination with the dual anti-HER2 blockade consisting of trastuzumab biosimilar ABP 980 and pertuzumab in early breast cancer patients with molecular HER2-enriched intrinsic subtype tested by PAM50.

DETAILED DESCRIPTION:
HER2-positive breast cancer is best defined by multiparameter gene expression profiling rather than analysis of the overexpression/amplification status of only HER2. As this subgroup is often correlated with a high expression of TILs and PD/PD-L1, immunogenic therapy strategies seem very promising. The pCR highly correlates with the overall outcome of patients with HER2-positive breast cancer [7]. Therefore, the pCR rate after neoadjuvant treatment has been adopted as a surrogate endpoint and, more recently, as a basis for accelerated drug approval [38].

Due to the high number of patients achieving a pCR after standard treatment of anti-HER2 therapy combined with chemotherapy, de-escalated strategies seem promising and designing a chemotherapy-free trial regimen is therefore modern, justifiable and of high scientific value. Therefore, we designed a prospective phase II, single arm, hypothesis-generating trial investigating the rate of pCR in patients with HER2-enriched breast cancer receiving four cycles of dual anti-HER2 blockade in combination with the checkpoint inhibitor pembrolizumab. Further translational research will be added to gain further insight into the tumor response or resistance to this treatment approach. The addition of standard chemotherapy after this study treatment will be at the discretion of the investigator. In case of a non-pCR after study treatment, continuing treatment with chemotherapy and antihormonal therapy in case of HR positive disease is highly recommended.

ELIGIBILITY:
Inclusion Criteria:

* Female participants, who are at least 18 years of age on the day of signing informed consent with newly histologically locally confirmed diagnosis of HER2neu 2+ or 3+ breast cancer.
* Have previously untreated, non-metastatic (M0) HER2-enriched breast cancer defined as the following combined primary tumor (T) and regional lymph node (N) staging per American Joint Committee on Cancer (AJCC) for breast cancer staging criteria version 7 as assessed by the Investigator based on radiological and/or clinical assessment:

T1c, N0-N2; T2, N0-N2; T3, N0-N2

* Patients with HER2-enriched, estrogen and/ or progesterone receptor positive or negative breast cancer defined by American Society of Clinical Oncology (ASCO) / College of American Pathologists (CAP) guidelines can be included.
* Availability of tumor imaging performed within three months prior to start of screening phase: breast ultrasound and computed tomography (CT) thorax/abdomen or chest X-ray/liver ultrasound, bone scan, mammography or breast magnetic resonance imaging (MRI) (according to local standard).
* Ability to provide archived tumor tissue sample or at least two newly obtained separate tumor cores from the primary tumor or excisional biopsy of a tumor lesion not previously irradiated at screening to the central laboratory. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred over slides. Newly obtained biopsies are preferred over archived tissue.

Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.

Patients are eligible to be included in the trial only if all of the following criteria apply [items 1-6 must be met by the patient to be enrolled into the trial and before the start of the screening phase]:

1. Female patients, who are at least 18 years of age on the day of signing informed consent, with newly histologically locally confirmed diagnosis of HER2neu 2+ or 3+ breast cancer.
2. Previously untreated, non-metastatic (M0) HER2-enriched breast cancer defined as the following combined primary tumor (T) and regional lymph node (N) staging per AJCC for breast cancer staging criteria version 7 as assessed by the investigator based on radiological and/or clinical assessment:

   * T1c, N0-N2;
   * T2, N0-N2;
   * T3, N0-N2.
3. Patients with HER2-enriched, estrogen and/or progesterone receptor-positive or -negative breast cancer defined by ASCO/CAP guidelines.
4. Availability of tumor imaging performed within three months prior to start of screening phase: breast ultrasound and CT thorax/abdomen or chest X-ray/liver ultrasound, bone scan, mammography or breast MRI (according to local standard).
5. Ability to provide an archived tumor tissue sample or at least two newly obtained separate tumor cores from the primary tumor or excisional biopsy of a tumor lesion not previously irradiated at screening to the central laboratory. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred over slides. Newly obtained biopsies are preferred over archived tissue.

   Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
6. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and if at least one of the following conditions applies:

   1. not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. a WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 7 months after the last dose of study treatment Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
7. The patient provides written informed consent for participation in the trial. The patient may also provide consent for future biomedical research. However, the patient may participate in the main trial without participating in future biomedical research.
8. Confirmed HER2neu (IHC 2+ status and amplification [e.g. by FISH] or IHC 3+ status) tumor identification by local pathology.
9. Confirmed HER2-enriched status by PAM50 testing.
10. Confirmed HR+ or HR- status.
11. Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or borderline, a serum pregnancy test will be required.

    Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for the patient to start receiving study medication.
12. Left ventricular ejection fraction (LVEF) of ≥55% or ≥ institution lower limit of normal (LLN) as assessed by echocardiogram (ECHO) or multigated acquisition (MUGA) scan performed at screening or performed in clinical routine within 6 weeks prior to first treatment allocation.
13. Normal ECG performed at screening or performed in clinical routine within 6 weeks prior to first treatment allocation.
14. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG performance status is to be performed within 10 days prior to the date of treatment initiation.
15. Adequate organ function as defined in the following table. Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

• Patients are excluded from the trial if any of the following criteria apply:

1. Patient has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T cell receptor (e.g. CTLA-4, OX 40, CD137) or has participated in MK-3475 clinical trials.
2. Patient has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to first dose of study medication.

   Note: Patients must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Patients with ≤Grade 2 neuropathy may be eligible.

   Note: If the patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
3. Patient has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.
4. Patient is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Patients who have entered the follow-up phase of an investigational trial may participate as long as it has been 4 weeks after the last dose of the previous investigational agent. Patient should be excluded if she received an investigational agent with anti-cancer or anti-proliferative intent within the last 12 months.
5. Patient has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
6. Prior malignancy with a disease-free survival of ≤5 years before signing informed consent.

   Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. ductal carcinoma in situ, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
7. Patient has a known hypersensitivity to the components of the study therapy, its analogs, murine proteins or any of the excipients.
8. Patient has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Patient has a significant cardiovascular disease, such as:

   * LVEF <55%
   * History of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the past 6 months
   * Congestive heart failure (CHF) New York Heart Association (NYHA) Class I-IV or history of CHF NYHA class III or IV
10. Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the trial, including but not confined to:

    * Unstable arrhythmias requiring treatment, i.e., atrial tachycardia with a heart rate ≥100/min at rest, significant ventricular arrhythmia (ventricular tachycardia) or higher-grade AV-block
    * Angina pectoris within the last 6 months requiring anti-anginal medication
    * Clinically significant valvular heart disease
    * Evidence of myocardial infarction on electrocardiogram (ECG)
    * Poorly controlled hypertension (e.g. systolic >180 mm Hg or diastolic >100 mm Hg).
11. Inadequate organ function including but not confined to:

    * hepatic impairment (Child Pugh Class C)
    * pulmonary disease (severe dyspnea at rest due to complications of advanced malignancy or requiring oxygen therapy).
12. Patient has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Patient has an active infection requiring systemic therapy.
14. Patient has a known history of human immunodeficiency virus (HIV), hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (defined as detectable HCV RNA [qualitative] is detected).

    Note: Testing of hepatitis B is required in all patients during screening as standard of care according to current guidelines in early breast cancer.

    HIV and hepatitis C testing is required in all patients with significant risk factors (see checklist below). There is a significant risk if one of the items on the checklist applies for the patient.
    * HIV and hepatitis C risk checklist:
    * Patient has frequently changing sexual partners.
    * Patient practices anal sex.
    * The patient has already been diagnosed with another sexually transmitted infection, such as syphilis or gonorrhea.
    * Patient suffers from drug abuse.
    * Tattoos or piercings abroad within the last 4 months.
    * Presence of a positive HIV and/or Hepatitis C test.
    * Patient received a blood transfusion before 1992.
    * Patient is an organ transplant recipient.
    * The patient's mother has/had HIV and/or hepatitis C.
    * Patient has elevated liver blood values (relevant for hepatitis C risk).
15. Patient has a known history of active TB (Bacillus Tuberculosis).
16. Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
17. Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Patient is pregnant or breastfeeding, or expecting to conceive children or planning to breastfeed within the projected duration of the trial, starting with the screening visit through 7 months after end of treatment.
19. Male patients with breast cancer.
20. History of breast cancer.
21. Factors indicating risk of poor compliance.
22. Pathological laboratory assessments:

    * Thrombocytopenia > CTCAE grade 1
    * Increases in ALT/AST > CTCAE grade 1
    * Hypokalemia > CTCAE grade 1
    * Neutropenia > CTCAE grade 1
    * Anemia > CTCAE grade 1
23. Non-operable breast cancer including inflammatory breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pCR rate of the combination therapy consisting of pembrolizumab in combination with the dual anti-HER2 blockade trastuzumab biosimilar ABP 980 and pertuzumab in patients with HER2-enriched early breast cancer assessed by PAM50 testing | After neoadjuvant treatment (planned duration of treatment is 12 weeks)
  pCR defined as no invasive tumor in breast and lymph nodes (ypT0/is, ypN0) at surgery after study treatment

SECONDARY OUTCOMES:
Number and percentage of fatal adverse events as assessed by CTCAE 5.0 | 9 months for individual participants
  AEs classified by System Organ Class (SOC) and Preferred Terms (PT), descriptive analysis by number of observations and their percentage.
Number and percentage of serious treatment-emergent adverse events as assessed by CTCAE 5.0 | 9 months for individual participants
  AEs classified by System Organ Class (SOC) and Preferred Terms (PT), descriptive analysis by number of observations and their percentage.
Number and percentage of treatment-related adverse events as assessed by CTCAE 5.0 | 9 months for individual participants
  AEs classified by System Organ Class (SOC) and Preferred Terms (PT), descriptive analysis by number of observations and their percentage.
Number and percentage of treatment-emergent adverse events of interest as assessed by CTCAE 5.0 | 9 months for individual participants
  AEs classified by System Organ Class (SOC) and Preferred Terms (PT), descriptive analysis by number of observations and their percentage.
Number and percentage of adverse events leading to investigational product discontinuation | 9 months for individual participants
  AEs classified by System Organ Class (SOC) and Preferred Terms (PT), descriptive analysis by number of observations and their percentage.
Number and percentage of severity of adverse events as assessed by CTCAE 5.0 | 9 months for individual participants
  Descriptive analysis by number of observations and their percentage.
Number and percentage of causality of adverse events as assessed by investigator and sponsor | 9 months for individual participants
  Descriptive analysis by number of observations and their percentage.
Number and percentage of outcome of adverse events as per investigator assessment | 9 months for individual participants
  Descriptive analysis by number of observations and their percentage.
Number and percentage of seriousness of adverse events as assessed by CTCAE 5.0 | 9 months for individual participants
  Descriptive analysis by number of observations and their percentage.

CONTACTS AND LOCATIONS:
Overall Officials: s.kuemmel@kem-med.com Kuemmel, Professor, Principal Investigator — Clinics Essen-Mitte, Breast Center
Locations (12):
- Germany (12):
  - Universitätsklinikum Tübingen Frauenklinik, Tübingen, Baden-Wurttemberg
  - Breast Center of the University of Munich (LMU) Universitätsfrauenklinik Großhadern, Munich, Bavaria
  - Rotkreuzklinikum München GmbH Frauenklinik, Munich, Bavaria
  - Niels-Stensen-Kliniken Franziskus-Hospital Harderberg Zentrum für Frauenheilkunde und Abteilung für Senologie, Georgsmarienhütte, Lower Saxony
  - Diakoniekrankenhaus Henriettenstiftung GmbH, Hanover, Lower Saxony
  - Onkologische Praxis, Bielefeld, North Rhine-Westphalia
  - St. Elisabeth Krankenhaus GmbH Brustzentrum, Cologne, North Rhine-Westphalia
  - Onkodok GmbH, Gütersloh, North Rhine-Westphalia
  - Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, North Rhine-Westphalia
  - Praxisnetzwerk, Troisdorf, North Rhine-Westphalia
  - Charité Campus Mitte Klinik für Gynäkologie, Berlin
  - Mammazentrum Hamburg, Hamburg

REFERENCES:
- [Derived] Kuemmel S, Graeser M, Schmid P, Reinisch M, Feuerhake F, Volk V, Armeanu-Ebinger S, Schutz L, Kelemen O, Schroeder C, Ossowski S, Jozwiak K, Kostara A, Scheffen I, Ludtke-Heckenkamp K, Hilpert F, Kentsch A, Ziske C, Depenbusch R, Braun M, Blohmer JU, Zu Eulenburg C, Christgen M, Bartels S, Kreipe HH, Wuerstlein R, Biehl C, Pelz E, Hartkopf A, Harbeck N, Gluz O; West German Study Group investigators. Chemotherapy-free neoadjuvant pembrolizumab combined with trastuzumab and pertuzumab in HER2-enriched early breast cancer (WSG-KEYRICHED-1): a single-arm, phase 2 trial. Lancet Oncol. 2025 May;26(5):629-640. doi: 10.1016/S1470-2045(25)00097-X. PMID 40318646